CLINICAL TRIAL: NCT03630770
Title: Effect of Medium Chain Triglyceride Intake on Colonization of Preterm Infants With Candida
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph Bliss (Other)
Collaborators: Tufts University (Other)
Responsible Party: Sponsor-Investigator, Joseph Bliss, Associate Professor of Pediatrics, Women and Infants Hospital of Rhode Island
Organization: Women and Infants Hospital of Rhode Island (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WIH 13-0088
Record Dates: First submitted 2018-07-25; First posted 2018-08-15 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Candida Infection; Premature Infant
MeSH Terms: conditions — Candidiasis; Premature Birth | interventions — Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group receives no feeding supplement.
- MCT Oil (Experimental): This group is supplemented with MCT oil
  Interventions: Drug: Medium-Chain Triglyceride (MCT) Oil

INTERVENTIONS:
Drug: Medium-Chain Triglyceride (MCT) Oil — Infants receive 0.5 ml/oz of MCT oil to their prescribed feedings for 21 days or until hospital discharge.
  Arms: MCT Oil

SUMMARY:
This study evaluates whether adding a dietary supplement similar to coconut oil (MCT oil) to feedings in premature infants will reduce the amount of yeast (Candida) detectable in their stool. Infants who have Candida in their stool are eligible to participate. Half of the enrolled infants will have additional MCT oil added to their feedings and half will not.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant admitted to the Neonatal Intensive Care Unit at Women & Infants Hospital
* Receiving full enteral feeds of either preterm or transitional formula or fortified breast milk
* Anticipated to have a minimum stay of two weeks

Exclusion Criteria:

* Prior exposure to antifungal drugs

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Bliss, MD, PhD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunsalus KT, Tornberg-Belanger SN, Matthan NR, Lichtenstein AH, Kumamoto CA. Manipulation of Host Diet To Reduce Gastrointestinal Colonization by the Opportunistic Pathogen Candida albicans. mSphere. 2015 Nov 18;1(1):e00020-15. doi: 10.1128/mSphere.00020-15. eCollection 2016 Jan-Feb. PMID 27303684
- [Result] Arsenault AB, Gunsalus KTW, Laforce-Nesbitt SS, Przystac L, DeAngelis EJ, Hurley ME, Vorel ES, Tucker R, Matthan NR, Lichtenstein AH, Kumamoto CA, Bliss JM. Dietary Supplementation With Medium-Chain Triglycerides Reduces Candida Gastrointestinal Colonization in Preterm Infants. Pediatr Infect Dis J. 2019 Feb;38(2):164-168. doi: 10.1097/INF.0000000000002042. PMID 29596218

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | MCT Oil
Started | 4 | 8
Completed | 4 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | MCT Oil | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Full Range); unit: weeks gestation] | 27.8 [23 to 32] | 25.5 [23 to 28] | 26.7 [23 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 5 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Maternal age [Mean (Standard Deviation); unit: years] | 29 (9) | 30 (10) | 29 (10)
Cesarean delivery [Count of Participants; unit: Participants] | 3 | 6 | 9
Prenatal steroids [Count of Participants; unit: Participants] | 3 | 6 | 9
Birth weight [Mean (Full Range); unit: grams] | 1032 [570 to 1490] | 745 [610 to 890] | 889 [570 to 1490]
Total parenteral nutrition duration [Mean (Full Range); unit: days] | 15.5 [4 to 40] | 16 [10 to 23] | 15.8 [4 to 40]
Umbilical line duration [Mean (Full Range); unit: days] | 4.5 [0 to 9] | 7.6 [4 to 13] | 6.1 [0 to 13]
Peripherally inserted central catheter duration [Mean (Full Range); unit: days] | 9.7 [0 to 32] | 7.6 [0 to 15] | 8.7 [0 to 32]
Breast milk feeds [Count of Participants; unit: Participants] | 3 | 5 | 8
Formula feeds [Count of Participants; unit: Participants] | 1 | 3 | 4
Postnatal steroids [Count of Participants; unit: Participants] | 0 | 3 | 3
Antacid treatment [Count of Participants; unit: Participants] | 0 | 0 | 0
Antibiotic duration [Mean (Full Range); unit: days] | 4.5 [0 to 7] | 8.1 [2 to 15] | 6.3 [0 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Stool Fungal Burden
Description: Change in colony-forming units (cfu) of Candida per gram of stool. Data table reflects total number of stool samples collected from subjects in each group that were included in the analysis.
Time Frame: Before supplementation, 1 week after supplementation begins, 3 weeks (at conclusion of supplementation)
Population: Candida colony counts per gram of stool in each sample
Measure: Median (Inter-Quartile Range); unit: cfu per gram
Units Other Than Participants: stool samples
Arm/Group | Control | MCT Oil
Number analyzed (Participants) | 4 | 8
Number analyzed (stool samples) | 50 | 130
cfu per gram
  Before supplementation: number analyzed (stool samples) | 11 | 21
  Before supplementation | 500 [26 to 21000] | 55000 [3885 to 86000]
  During supplementation: number analyzed (stool samples) | 20 | 50
  During supplementation | 1671 [42.5 to 108500] | 622.5 [43 to 3925]
  After supplementation: number analyzed (stool samples) | 19 | 59
  After supplementation | 1744 [23 to 26330] | 2364 [800 to 7000]
Statistical Analysis 1: Comparison: Control; Stool fungal counts (cfu/g) were compared between groups using negative binomial regression within time period (before, during, after). Rate ratio was calculated to reflect the direction and magnitude of change in stool colony counts between time periods (before v. during supplementation) for the control group; Test type: Other; p = 0.9, Negative binomial regression — p-values underwent generalized estimating equations adjustment for multiple measures per individuals within time; Rate Ratio = 0.98, 95% CI 2-sided [0.55 to 1.7]
Statistical Analysis 2: Comparison: Control; Stool fungal counts (cfu/g) were compared between groups using negative binomial regression within time period (before, during, after). Rate ratio was calculated to reflect the direction and magnitude of change in stool colony counts between time periods (during v. after supplementation) for the control group; Test type: Other; p < 0.001, Negative binomial regression — p-values underwent generalized estimating equations adjustment for multiple measures per individuals within time; Rate Ratio = 8.1, 95% CI 2-sided [2.6 to 25]
Statistical Analysis 3: Comparison: MCT Oil; Stool fungal counts (cfu/g) were compared between groups using negative binomial regression within time period (before, during, after). Rate ratio was calculated to reflect the direction and magnitude of change in stool colony counts between time periods (before v. during supplementation) for the MCT group; Test type: Other; p = 0.02, Negative binomial regression — p-values underwent generalized estimating equations adjustment for multiple measures per individuals within time; Rate Ratio = 0.15, 95% CI 2-sided [0.03 to 0.75]
Statistical Analysis 4: Comparison: MCT Oil; Stool fungal counts (cfu/g) were compared between groups using negative binomial regression within time period (before, during, after). Rate ratio was calculated to reflect the direction and magnitude of change in stool colony counts between time periods (during v. after supplementation) for the MCT group; Test type: Other; p < 0.001, Negative binomial regression — p-values underwent generalized estimating equations adjustment for multiple measures per individuals within time; Rate Ratio = 61, 95% CI 2-sided [6.9 to 533]

ADVERSE EVENTS:
Time Frame: Through duration of hospitalization, an average of 3 weeks
Arm/Group | Control | MCT Oil
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03630770/Prot_000.pdf